CLINICAL TRIAL: NCT05069402
Title: Impact of Immunomodulating Oral Nutrition on Surgical Complications
Brief Title: Impact of Various Diets on Surgical Complications
Acronym: IMM4
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanley Dudrick's Memorial Hospital (Other)
Responsible Party: Principal Investigator, Stanislaw Klek, Head of the Unit, Stanley Dudrick's Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 4armsimmuno
Record Dates: First submitted 2021-09-25; First posted 2021-10-06 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2021-10

CONDITIONS: Complication,Postoperative
MeSH Terms: conditions — Postoperative Complications | interventions — Immunonutrition Diet

STUDY DESIGN:
Intervention Model Description: randomisation into 4 arms
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The physician is unaware of the type of the intervention. The type of intervention is given by the independent person to dietitian instructing the patient how to use the product.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Immunonutrition (Experimental): Oral immunonutrition containing arginine, omega-PUFAs and antioxidants
  Interventions: Dietary Supplement: Immunonutrition
- High-protein diet (Active Comparator): Oral nutrition with high-protein content
  Interventions: Dietary Supplement: High-protein
- Standard nutrition (Active Comparator): Oral nutrition with standard components
  Interventions: Dietary Supplement: Standard ONS

INTERVENTIONS:
Dietary Supplement: Immunonutrition — diet with immunonutrients
  Arms: Immunonutrition
Dietary Supplement: High-protein — Oral nutrition with high-protein content
  Arms: High-protein diet
Dietary Supplement: Standard ONS — Oral nutrition with standard ingredients
  Arms: Standard nutrition

SUMMARY:
The optimalisation of the health status of patients scheduled for major surgery has been considered to be the most important point of perioperative care, and nutritional intervention has been perceived a key point of that intervention. Immunomodulating diets were thought to reduce cmplications, hoever recent studies put that opnion in doubt. This study was designed to assess the actual clinical significance of oral immunonutrition.

DETAILED DESCRIPTION:
The optimalisation of the health status of patients scheduled for major surgery has been considered to be the most important point of perioperative care, and nutritional intervention has been perceived a key point of that intervention. Italian studies followed by metanalyses demonstrated the superiority of immunomodulating diets (IM) over any other preoperative nutrition, hence the surgical guidelines for enteral nutrition published by European Society for Clinical Nutrition and Metabolism (ESPEN) in 2006 recommended to use IM for 7-14 days preoperatively in all patients undergoing major surgeries. Some authors questioned IM by showing no benefit of IM over standard enteral nutrition. Other authors observed similar results.The debate was far from being over - in 2015 a new metanalysis stated that perioperative enteral nutrition is the best option for managing clinical status of patients who underwent selective surgery for gastrointestinal cancer. One year later, ESPEN changed its surgical recommendations and advised to use IM preoperatively in malnourished and perioperatively in well-nourished patients. American recommendations remained unchanged and, according to them, it is advised to use IM preoperatively in all surgical patients, however, high-protein nutrition could also be an beneficial option.

To address those doubts and to assess the actual clinical significance of oral immunonutrition, a randomized, two center, prospective clinical trial was conducted.

ELIGIBILITY:
Inclusion Criteria:

* no sign of malnutrition (defined as one of the following unintentional weight loss by at least 10% or body mass index (BMI) < 18),
* good general status (Karnofsky Performance Index > 80,
* Eastern Cooperative Oncology Group (ECOG) grade 0 or 1);
* no confirmed neoplastic dissemination no severe concomitant disease (heart, lung, kidney, liver failure, chronic obstructive pulmonary disease [COPD], coronary aortic bypass graft [CABG], etc.),
* no history of known allergies or drug intolerance to analyzed substances.

Exclusion Criteria:

* Patients malnourished or with metastatic disease,
* pregnant,
* in poor general status (Karnofsky <80, Eastern Cooperative Oncology Group (ECOG) > 1),
* recent history of severe heart, lung, kidney or liver failure,
* history of allergies or drug intolerance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Surgical complications | 6 months
  Number and type of surgical complications
Infectious complications | 6 months
  Number and type of infectious complications

SECONDARY OUTCOMES:
Length of stay | 6 months
  Days of hospital stay after the operation

CONTACTS AND LOCATIONS:
Overall Officials: Stanislaw Klek, PhD, Principal Investigator — Stanley Dudrick's Memorial Hospital
Locations (2):
- Poland (2):
  - Narodowy Instytut Onkologii, Krakow, Malopolska
  - Stanley Dudrick's Memorial Hospital, Skawina, Malopolska

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR
Time Frame: 12 months
Access Criteria: any health professional